CLINICAL TRIAL: NCT04014881
Title: Single-center, Open-label, Single-arm Clinical Study of Efficacy and Safety of Anti-CD123 CAR-T Therapy in Patients With Refractory/Relapsed CD123+ Acute Myeloid Leukemia.
Brief Title: Safety and Efficacy of Anti-CD123 CAR-T Therapy in Patients With Refractory/ Relapsed CD123+ Acute Myeloid Leukemia.
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Collaborators: Wuhan Bio-Raid Biotechnology Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, MEI HENG, Principal Investigator, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WHUH-CART-CD123-01
Record Dates: First submitted 2019-07-02; First posted 2019-07-10 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: CD123+ Acute Myeloid Leukemia

STUDY DESIGN:
Intervention Model Description: This study was a single-center, open-label, single-arm, non-randomized,3+3 dose escalation clinical trial.Each dose group has 3 patients.If no DLT emerges in the group, then the next group uses the subsequent higher dose. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level. The maximum dose could be extended.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CD123+ Acute Myeloid Leukemia (Experimental): Patients will receive CD123-targeted CAR-T cells in the dose-climbing trial. Each dose group has 3 patients and the the maximum dose can be extended.
  Interventions: Biological: Third-generation anti-CD123 CAR-T cells

INTERVENTIONS:
Biological: Third-generation anti-CD123 CAR-T cells — From the minimum dose, If no DLT emerges in the group, then the next group uses the subsequent higher dose. If DLT emerges in a single subject in any dose level, 3 more subjects will be enrolled to the same dose level.

SUMMARY:
This is a single-center, open-label, single-arm study to evaluate the safety and efficacy of anti-CD123 CAR-T cells in patients with refractory/relapsed CD123+ Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
CD123 is a transmembrane subunit of the IL-3 receptor expressed on AML blasts. The investigators have conducted a third generationCD123-targeted CAR containing CD137 and CD28 costimulatory domains.This study aims to evaluate the safety and efficacy of anti-CD123 CAR-T cells in patients with relapsed/refractory CD123+ Acute Myeloid Leukemia.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological and histological examination confirmed CD123+ refractory or relapsed Acute Myeloid Leukemia.

   A. Diagnostic criteria for recurrent AML: After complete remission (CR), leukemia cells or bone marrow primordial cells > 0.050 (except for bone marrow regeneration after consolidation chemotherapy) or extramedullary leukemia cell infiltration appears again in peripheral blood.

   B．Diagnostic criteria for refractory AML(Meeting one of the following)

   i. ineffectiveness after the first standard regimen treatment of 2 courses.

   ii. patients relapse within 12 months after consolidation and intensive treatment after CR.

   iii. Patients relapse 12 months later and fail to respond to conventional chemotherapy.

   iv. Patients with two or more recurrences.

   v. Patients with persistent extramedullary leukemia.

   vi. Patients with recurrence after CR and unsuitable for HSCT (auto/allo-HSCT).
2. Aged 18 to 70 years (including 18 and 70 years old).
3. At least one measurable or evaluable lesion：AML patients with positive or relapsed positive bone marrow MRD.
4. ECOG≤ 2 and expected lifetime ≥3 months.
5. Adequate organ function:

   A. Liver function: ALT/AST≤3 ULN. Total bilirubin≤2 ULN.

   B. Renal function: eGFR> 60 mL/min/1.73 m2, or creatinine clearance ≥45mL/min.

   C. Lung function: Carbon Monoxide (DLCO) or Forced Expiratory Volume in the first second (FEV1) > 45% predicted.

   D. Cardiac function: LVEF ≥ 50%.
6. The patients did not receive any anticancer treatments such as chemotherapy, radiotherapy and immunotherapy (such as immunosuppressive drugs) within 4 weeks before admission, and the toxicity related to previous treatments had returned to < 1 level at admission (except for low toxicity such as alopecia).
7. Women of child-bearing potential and all male participants must use effective methods of contraception for at least 12 months after infusion.
8. Informed Consent/Assent: All subjects must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

1. Women who are pregnant (urine/blood pregnancy test positive) or lactating.
2. Male or female with a conception plan in the past 1 years.
3. Patients cannot guarantee effective contraception (condom or contraceptives, etc.) within 1 years after enrollment.
4. Uncontrolled infectious disease within 4 weeks prior to enrollment.
5. Active hepatitis B/C virus.
6. HIV infected patients.
7. Suffering from a serious autoimmune disease or immunodeficiency disease.
8. The patient is allergic and is allergic to macromolecular biopharmaceuticals such as antibodies or cytokines.
9. The patient participated in other clinical trials within 6 weeks prior to enrollment.
10. Systemic use of hormones within 4 weeks prior to enrollment (except for patients with inhaled corticosteroids).
11. Suffering from mental illness.
12. Patient has drug abuse/addiction.
13. Central nervous system involvement.
14. According to the investigator's judgment, the patient has other unsuitable grouping conditions.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-07-06 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-related Adverse Events | 3 years
  Therapy-related adverse events will be recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 4.0).

SECONDARY OUTCOMES:
Overall remission rate(ORR) of anti-CD123 CAR-T Therapy in patients with refractory/relapsed CD123+ Acute Myeloid Leukemia | 3 years
  ORR will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
Overall survival(OS) of anti-CD123 CAR-T cells in patients with refractory/relapsed CD123+ Acute Myeloid Leukemia | 3 years
  OS will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
Duration of Response(DOR) of anti-CD123 CAR-T cells in patients with refractory/relapsed CD123+ Acute Myeloid Leukemia | 3 years
  DOR will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
Progress-free survival(PFS) of anti-CD123 CAR-T cells in patients with refractory/relapsed CD123+ Acute Myeloid Leukemia | 3 years
  PFS will be assessed from the first CAR-T cell infusion to death or last follow-up (censored).
Rate of anti-CD123 CAR-T cells in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) rate and quantity of anti-CD123 CAR-T cells were determined by means of flow cytometry.
Quantity of anti-CD123 CAR copies in bone marrow cells and peripheral blood cells | 3 years
  In vivo (bone marrow and peripheral blood) quantity of anti-CD123 CAR copies were determined by means of qPCR.

CONTACTS AND LOCATIONS:
Overall Officials: Heng Mei, M.D., Ph.D, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

REFERENCES:
- [Background] Hansrivijit P, Gale RP, Barrett J, Ciurea SO. Cellular therapy for acute myeloid Leukemia - Current status and future prospects. Blood Rev. 2019 Sep;37:100578. doi: 10.1016/j.blre.2019.05.002. Epub 2019 May 11. PMID 31109711
- [Background] Arcangeli S, Rotiroti MC, Bardelli M, Simonelli L, Magnani CF, Biondi A, Biagi E, Tettamanti S, Varani L. Balance of Anti-CD123 Chimeric Antigen Receptor Binding Affinity and Density for the Targeting of Acute Myeloid Leukemia. Mol Ther. 2017 Aug 2;25(8):1933-1945. doi: 10.1016/j.ymthe.2017.04.017. Epub 2017 May 4. PMID 28479045
- [Background] Cartellieri M, Feldmann A, Koristka S, Arndt C, Loff S, Ehninger A, von Bonin M, Bejestani EP, Ehninger G, Bachmann MP. Switching CAR T cells on and off: a novel modular platform for retargeting of T cells to AML blasts. Blood Cancer J. 2016 Aug 12;6(8):e458. doi: 10.1038/bcj.2016.61. PMID 27518241
- [Background] Tettamanti S, Biondi A, Biagi E, Bonnet D. CD123 AML targeting by chimeric antigen receptors: A novel magic bullet for AML therapeutics? Oncoimmunology. 2014 May 14;3:e28835. doi: 10.4161/onci.28835. eCollection 2014. PMID 25083319
- [Background] Tasian SK, Kenderian SS, Shen F, Ruella M, Shestova O, Kozlowski M, Li Y, Schrank-Hacker A, Morrissette JJD, Carroll M, June CH, Grupp SA, Gill S. Optimized depletion of chimeric antigen receptor T cells in murine xenograft models of human acute myeloid leukemia. Blood. 2017 Apr 27;129(17):2395-2407. doi: 10.1182/blood-2016-08-736041. Epub 2017 Feb 28. PMID 28246194
- [Background] Mardiros A, Dos Santos C, McDonald T, Brown CE, Wang X, Budde LE, Hoffman L, Aguilar B, Chang WC, Bretzlaff W, Chang B, Jonnalagadda M, Starr R, Ostberg JR, Jensen MC, Bhatia R, Forman SJ. T cells expressing CD123-specific chimeric antigen receptors exhibit specific cytolytic effector functions and antitumor effects against human acute myeloid leukemia. Blood. 2013 Oct 31;122(18):3138-48. doi: 10.1182/blood-2012-12-474056. Epub 2013 Sep 12. PMID 24030378